CLINICAL TRIAL: NCT04480450
Title: Rituximab in Chronic Inflammatory Demyelinating Polyneuropathy: A Phase II Study
Brief Title: Rituximab in Chronic Inflammatory Demyelinating Polyneuropathy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to acquire funding
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R4CIDP
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Chronic Inflammatory Demyelinating Polyneuropathy
Keywords: CIDP
MeSH Terms: conditions — Polyradiculoneuropathy, Chronic Inflammatory Demyelinating | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- IVIg/SCIg < 3 Years Arm (Active Comparator): Patients with CIDP successfully treated with IVIg/SCIg for under 12 months. Subjects will receive an intravenous infusion of 1,000mg Rituximab at Week 0 and Week 2.
  Interventions: Drug: Rituximab
- IVIg/SCIg > 3 Years Arm (Active Comparator): Patients with CIDP successfully treated with IVIg/SCIg for more than 12 months. Subjects will receive an intravenous infusion of 1,000mg Rituximab at Week 0 and Week 2.
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Rituximab is a highly purified, 1328-amino acid antibody with an approximate molecular mass of 145 kD. Rituximab is a mouse human chimeric monoclonal antibody against CD20. Administration leads to between 90 and 100% peripheral B cell depletion via complement dependent cytotoxicity.

SUMMARY:
CIDP is a heterogeneous disease with variable responses to therapy. Recently, a distinctive subgroup of patients with serum autoantibodies to the paranodal proteins contactin and neurofascin have been identified. Although they present with active and serious disease, multiple clinical reports suggest that these patients can be cured with a treatment that depletes B cells and presumably eliminates pathogenic autoantibodies. However, beyond that subgroup of CIDP patients, which CIDP patients might benefit from Rituximab and B cell depletion is unknown. This Phase II study will treat 3 homogenous groups of 16 CIDP patients each with Rituximab in order to determine if there are subgroups that can be taken off current medications and put into long-term remission. The results from this study will be used to design a future larger trial. Biomarkers including paranodal antibodies, serum neurofilament light chains, anti-ganglioside antibodies will be obtained in order to learn about disease pathogenesis and possibly target therapy

ELIGIBILITY:
INCLUSION CRITERIA

1. Written informed consent obtained from subjects indicating that they understand the purpose of and procedures required for the study and are willing to participate
2. Male or female, aged ≥18 years
3. Documented diagnosis of typical CIDP according to the European Academy of Neurology/Peripheral Nerve Society criteria 202127
4. Must be willing to complete the study and return for follow-up visits.
5. Men and women of reproductive potential must agree to use an acceptable method of birth control during treatment and for twelve months (1 year) after completion of treatment.
6. Successfully treated CIDP patients. Data at or prior to the screening visit must show evidence that during the course of therapy either the INCAT score improved by 1 or more points or improvement occurred according to the physician opinion.
7. CIDP disease stability is based on 2 visits that are 3 or more months apart documented at or prior to the screening visit by assessing unchanged CIDP status per physician opinion. The subject must be at the same dosage and frequency of CIDP therapy in between these 2 timepoints.
8. Belonging to 1 of the following 2 treatment groups:

   1. IVIg/SCIg for up to 3 years.
   2. IVIg/SCIg for more than 3 years.
9. Off steroids for at least 3 months before screen visit. Topical steroids and infrequent intraarticular steroids are allowed.
10. No anticipated change in dosage or CIDP therapy from week 0 to week 24.
11. Off concurrent immunosuppressive agents (such as azathioprine, methotrexate, mycophenolate mofetil, or cyclosporine or cyclophosphamide or any other agent) for at least 6 months prior to screening visit.

EXCLUSION CRITERIA

1. Female subjects who are premenopausal and are

   1. pregnant on the basis of a serum pregnancy test,
   2. breast-feeding, or
   3. not using an effective method of double barrier (1 hormonal plus 1 barrier method or 2 simultaneous barrier methods) or birth control (birth control pills, male condom, female condom, intrauterine device, Norplant, tubal ligation, or other sterilization procedures).
2. Participation in another clinical study within 30 days before entering the study or during the study
3. Employee or direct relative of an employee of the study site or Sponsor
4. Other medical condition, laboratory finding, or physical exam finding that precludes participation
5. A neuropathy of other causes, including:

   1. A motor syndrome that fulfils criteria for multifocal motor neuropathy (MMN) with conduction block
   2. CIDP with monoclonal gammopathy of uncertain significance (CIDP-MGUS) or monoclonal gammopathy associated with an oncologic diagnosis
   3. Neuropathies secondary to infections, disorders, or systemic diseases
   4. Drug-, biologic-, chemotherapy-, or toxin-induced peripheral neuropathy
   5. Hereditary demyelinating neuropathies
   6. Central demyelinating disorders (e.g. multiple sclerosis)
   7. Others, like polyneuropathy, lumbosacral radiculoplexus neuropathy
6. Patients with known history prior to screening visit of nodal and paranodal (anti-NF155, anti- CNTN1, anti- Caspr1 or anti-NF140/186 antibody) performed at a laboratory meeting quality standards for cell-based assay method and if required other confirmatory assays
7. Any chronic or debilitating disease, or central nervous disorder that causes neurological symptoms or may interfere with assessment of CIDP or outcome measures
8. Cardiac insufficiency (New York Heart Association Classes III/IV), cardiomyopathy, significant cardiac arrhythmia requiring treatment, unstable or advanced ischemic heart disease, congestive heart failure or severe hypertension
9. Subjects with current malignancy requiring chemotherapy and/or radiotherapy, or history of malignancy with less than 2 years of complete remission prior to screening. Exceptions are: adequately treated basal cell or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, and stable prostate cancer not requiring treatment
10. Plasma exchange within the last 3 months of screen visit.
11. Any prior treatment with a biologic (e.g. rituximab (MabThera®/Rituximab®), ocrelizumab (Ocrevus®), natalizumab (Tysabri®), alemtuzumab, TNF-α inhibitor)
12. Abnormal laboratory parameters:

    1. creatinine >1.5 times the upper normal limit (UNL)
    2. hemoglobin (Hb) <10 g/dL
    3. absolute neutrophil count (ANC) <1000 cells/μl
    4. elevated liver enzymes (AST or ALT >2.5 x Upper Limit of Normal).
    5. platelets < 100,000/mL
13. History of bone marrow hypoplasia, leucopenia, thrombocytopenia, significant anemia, clinical or laboratory evidence of immunodeficiency syndromes, that are not transient events or side effects related to a clinical procedure (i.e. plasmapheresis) and within one year of screening.
14. Positive Hepatitis B or C serology (Hep B surface antigen and Hep C antibody). For patients who are negative for surface antigen [HBsAg] and positive for HB core antibody [HBcAb+], we will consult liver disease experts before starting and during treatment
15. History of positive HIV (HIV conducted during screening if applicable)
16. Receipt of a live vaccine within 4 weeks prior to randomization
17. Contraindication to receiving rituximab
18. History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
19. History of recurrent significant infection or history of recurrent bacterial infections
20. Known active bacterial, viral fungal mycobacterial, or other infection (including tuberculosis or atypical mycobacterial disease, but excluding fungal infections of nail beds) or any major episode of infection requiring hospitalization or treatment with IV antibiotics within 4 weeks of screening or oral antibiotics within 2 weeks prior to screening
21. Lack of venous access
22. History of drug, alcohol, or chemical abuse within 6 months prior to screening
23. Any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the subject at high risk from treatment complications
24. Levels of IgG or IgM that are below 30% of the lower limit of normal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-07 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Inflammatory Neuropathy Cause and Treatment (INCAT) Disability Score | 48 Weeks
  The INCAT disability scale captures upper and lower limb dysfunction separately on a scale of 0 to 5, which are then added together for a total composite score ranging between 0 and 10.15 Lower scores indicate no or minimal disability (no arm dysfunction or walking abnormality), and higher scores indicate more disability (no purposeful arm movement or restricted to wheelchair). The adjusted INCAT disability score is identical to the INCAT disability score with the exception that changes in upper limb function from 0 (normal) to 1 (minor symptoms) are excluded. This exclusion was made because upper limb changes from 0 to 1 (minor symptoms in the fingers which do not impair any functional activities) were not judged by regulatory agencies to be clinically significant in all patients. With the exception of a change in the upper limb score from 0 to 1, all other 1 point changes in the INCAT score are considered clinically significant.

SECONDARY OUTCOMES:
Inflammatory-Rasch-built Overall Disability Scale (I-RODS) | 48 Weeks
  The Rasch built overall disability scale for immune-mediated peripheral neuropathies (I-RODS) is a patient-based, linearly weighted scale that captures activity and social participation limitations in patients with CIDP.16 The assessment includes 24 questions that address upper and lower limb disability. These range in difficulty from ability to read a book, eat, or brush teeth to dance, stand for hours, and run. Participants are asked to indicate if they can easily perform the task, perform it with difficulty, or are unable to perform it at all. Both the ability of the patient and the perceived difficulty of a task are tallied for a raw R-ODS score that ranges between 0 (complete disability) and 48 (no disability). The resulting raw I-RODS score are then be transformed to a final I-RODS score ranging from 0 (severe disability) to 100 (no disability). A change in the I-RODS scores of ≥ 4 points (using the centile metric) is considered clinically meaningful.
Modified Fatigue Severity Scale (mFSS) | 48 Weeks
  The fatigue severity scale (FSS) is one available tool to measure fatigue.17 FSS is a Rasch-built patient self-assessment questionnaire that measures fatigue severity and impact on activities and lifestyle by asking participants to respond to 7 separate items. Responses are scored on a 4-point scale (0= strongly disagree, 3 = strongly agree) with a total score range from 0 to 21. Higher scores indicate more fatigue.
Visual Analog Pain Severity Scale (VAS) | 48 Weeks
  The pain VAS is a validated sensitive linear scale that has been widely used to assess pain in diverse populations of patients.18 The scale is comprised of a horizontal or vertical line, 10 centimeters in length, anchored by 2 verbal descriptors, one for each symptom extreme. A score of 0 indicates "no pain" while a score of 100 (100 mm scale) indicates "pain as bad as it could be" or "worst imaginable pain". The pain VAS is self-completed by the respondent by placing a line perpendicular to the VAS line at the point that represents their pain intensity. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. Higher scores indicate greater pain intensity
Martin vigorimeter grip strength | 48 Weeks
  Grip strength provides a quantitative objective measure of grip strength and an instant measure of strength impairment. The Vigorimeter from Martin is a hand-held device that measures grip strength by recording the pressure generated from squeezing a rubber bulb. The rubber bulb is placed in the hand between the palm and the thumb and index fingers. Pressure expressed in Kilopascal is recorded with a nanometer. A result is obtained after the subject squeezes 3 times with each hand. The mean grip strength of three squeezes is recorded in each hand.
Medical Research Council (MRC) Sum Score | 48 Weeks
  The MRC sum score is determined by assessing the following 8 muscle pairs: bilateral shoulder abduction, elbow flexion, wrist extension, hip flexion, knee extension, index finger abduction, great toe dorsiflexion and foot dorsiflexion. The MRC sum score is a summation of the MRC grades (range 0 to 5 with 0 = paralysis; 1 = only a trace or flicker of muscle contraction is seen or felt; 2 = muscle movement is possible with gravity eliminated; 3 = muscle movement is possible against gravity; 4 = muscle strength is reduced, but movement against resistance is possible and 5 = normal strength given in full numbers. The MRC sum score ranges from 0 ("total paralysis") to 60 ("normal strength").
EuroQOL-5D | 48 Weeks
  The EuroQOL-5D is a simple survey meant to assess quality of life in a wide range of health conditions.23 The measure has 2 parts. In the first part 5 health dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) are assessed by 1 of 5 levels of impairment: no problems, slight problems, moderate problems, severe problems, or extreme problems. The second part of the survey is a visual analogue scale assessing overall health on the day of assessment. The EuroQOL-5D has been extensively validated in numerous therapeutic areas and has been found to be sensitive, reliable, and have good internal consistency.

CONTACTS AND LOCATIONS:
Overall Officials: Mazen Dimachkie, MD, Principal Investigator — University of Kansas Medical Center

IPD SHARING:
Plan to Share IPD: Undecided